CLINICAL TRIAL: NCT06843057
Title: Effectiveness of Kinesiotaping Along with Mulligan's Mobilization with Movement on Improving Pain and Function in Patients with Adhesive Capsulitis of Shoulder: a Randomized Controlled Trial
Brief Title: Kinesiotaping Along with Mulligan's Mobilization with Movement in Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AWH/EC/03/2021/3
Record Dates: First submitted 2025-02-15; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Adhesive Capsulitis
Keywords: Rehabilitation; Manual Therapy; Exercise Therapy; Shoulder Pain
MeSH Terms: conditions — Bursitis; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Two Parallel Arms Experimental Design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group received Kinesiotaping, Mulligan's mobilization with movement, and conventional physiotherapy.
  Interventions: Other: Kinesio taping; Other: Mulligan's mobilization with movement techniques; Other: Conventional physiotherapy
- Control Group (Active Comparator): Control group received only Mulligan's mobilization with movement and conventional physiotherapy
  Interventions: Other: Mulligan's mobilization with movement techniques; Other: Conventional physiotherapy

INTERVENTIONS:
Other: Kinesio taping — Kinesio taping is a therapeutic technique that involves applying a special elastic tape to the skin to support and stabilize muscles and joints without restricting their range of motion.
  Arms: Experimental Group
Other: Mulligan's mobilization with movement techniques — Mulligan's mobilization with movement (MWM) techniques involve the application of a sustained manual force or glide to a joint while the patient actively performs a movement that is typically painful or restricted.
Other: Conventional physiotherapy — Mulligan Mobilization with Movement, Ultrasound Therapy, Active assisted ROM exercises for shoulder, Capsular Stretching exercises

SUMMARY:
The study aimed to evaluate the effectiveness of combining Kinesiotaping with Mulligan's mobilization with movement in treating shoulder adhesive capsulitis. Thirty patients participated in a randomized control trial, divided equally into an experimental group and a control group. The experimental group received Kinesiotaping, Mulligan's mobilization with movement, and conventional physiotherapy, while the control group received only Mulligan's mobilization with movement and conventional physiotherapy. Pain, range of motion, and functional outcomes were measured using a visual analogue scale, goniometer, and the Shoulder Pain and Disability Index (SPADI) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Primary adhesive capsulitis,
* Controlled diabetes mellitus,
* Restriction of movements in capsular pattern,
* Shoulder pain for more than one month.

Exclusion Criteria:

* Secondary adhesive capsulitis,
* Cancer,
* Bilateral adhesive capsulitis,
* Skin infections in the shoulder region,
* Shoulder joint infections,
* Wounds or ulcers in the shoulder region,
* Hypersensitivity to tape,
* Recent shoulder dislocation,
* Recent shoulder fractures.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | From enrollment to the end of treatment at 4 weeks
  The Visual Analog Scale (VAS) is a tool for measuring subjective experiences, like pain. It's typically a 10 cm line, with endpoints marking the extremes (e.g., "no pain" to "worst imaginable pain"). The minimum value is 0, and the maximum is 10. Respondents mark a point on the line that corresponds to their experience. Higher scores usually indicate worse outcomes for negative experiences like pain.
Range of motion | From enrollment to the end of treatment at 4 weeks
  Range of motion (ROM) measures the movement extent of a joint or body part, expressed in degrees. Minimum values indicate restricted movement (e.g., 0° signifies no movement), while maximum values represent full movement capacity (e.g., 180° for shoulder flexion). Higher scores generally indicate a better outcome, as they reflect greater flexibility and joint function.
Shoulder Pain and Disability Index | From enrollment to the end of treatment at 4 weeks
  The Shoulder Pain and Disability Index (SPADI) is a 13-item questionnaire assessing pain and disability due to shoulder issues. Scores range from 0 to 100, with 0 indicating no pain/disability and 100 indicating severe pain/disability. Higher scores signify worse outcomes, reflecting greater pain and functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, MPTh, Principal Investigator — King Saud University
Locations (1):
- AWH Special College, Calicut, Kerala, India

IPD SHARING:
Plan to Share IPD: No